CLINICAL TRIAL: NCT01849081
Title: Evaluating the Efficacy of CPAP Therapy for the Treatment of Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Evaluating the Efficacy of CPAP Therapy for the Treatment of Fatty Liver
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in priorities, study closed prior to enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kathleen E Corey, Instructor in Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000688
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; Obstructive sleep apnea
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CPAP (Experimental): Subjects in this arm with receive treatment with CPAP for fatty liver disease.
  Interventions: Device: CPAP
- Lifestyle Intervention (Active Comparator): Subjects in the lifestyle arm will undergo 12 weeks of dietary counseling.
  Interventions: Behavioral: LIfestyle

INTERVENTIONS:
Device: CPAP — Subjects in the intervention arm will be treated with continuous positive airway pressure (CPAP) device at night.
  Arms: CPAP
Behavioral: LIfestyle — Subjects will undergo 12 weeks of dietary counseling.
  Arms: Lifestyle Intervention

SUMMARY:
We are doing this research study to evaluate whether continuous positive airway pressure (CPAP), a treatment for sleep apnea, will also help treat fatty liver disease. Sleep apnea is a disease where a person has interruptions in their breathing while they are sleep. This can lead to low oxygen levels in the blood. CPAP is a mask that delivers oxygen at high pressure to the lungs to prevent a decrease in blood oxygen levels. CPAP is a known treatment for sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older with a previous liver biopsy showing NASH and at least grade 2 steatosis
* Obstructive sleep apnea diagnosed by sleep study.

Exclusion Criteria:

* Other causes of chronic liver disease
* cirrhosis
* less than 33% steatosis identified on magnetic resonance spectroscopy (MRS)
* Alcohol use >2 units per day for women or >3 units per day for men
* Intolerance to or refusal of CPAP therapy
* overnight desaturation (more than 10% of the sleep time with oxygen desaturation below 85%)
* underlying sever sleepiness (Epworth scale more than 15)
* uncontrolled hypertension
* Severe heart failure (ejection fracture less than 30%)
* cardiac arrhythmias (atrial fibrillation or history of ventricular tachycardia)
* those who are commercial drivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Steatosis by MRS | 12 weeks
  Subjects will undergo baseline and 12 week magnetic resonance spectroscopy to assess the impact of CPAP or diet on fatty liver.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen E Corey, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States